CLINICAL TRIAL: NCT03073408
Title: Design of a Closed-loop Controller for the Administration of Propofol Based on the Bispectral Index (BIS). Effectiveness of the Smith Predictor and Comparison With Manual Control
Brief Title: Design of a Closed-loop Controller Based on the Bispectral Index (BIS) Effectiveness of the Smith Predictor
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: José Antonio Reboso Morales (Other)
Collaborators: University of La Laguna (Other)
Responsible Party: Sponsor-Investigator, José Antonio Reboso Morales, MD, PhD, Hospital Universitario de Canarias
Organization: Hospital Universitario de Canarias (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2017_
Record Dates: First submitted 2017-02-24; First posted 2017-03-08 (Actual); Last update posted 2017-03-08 (Actual); Status verified 2017-03

CONDITIONS: General Anesthesia
Keywords: Propofol; Bispectral index (BIS); Closed loop
MeSH Terms: interventions — Propofol

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1: Manual control group (Active Comparator): The propofol infusion rate is adjusted manually in a pump by the investigator to maintain BIS between 40 and 60. For this titration it is necessary continuous monitoring, clinical experience, and pharmacokinetic/pharmacodynamic knowledge.
  Interventions: Drug: Propofol
- 2: PI +Smith group (Experimental): The closed loop control automatically adjust propofol infusion rate guided by the feedback of the real value of BIS. The automatic system has to achieve a target BIS of 50 and maintain it between 40 and 60.
  Interventions: Drug: Propofol

INTERVENTIONS:
Drug: Propofol — Closed loop control for propofol administration guided by the BIS.
  Arms: 2: PI +Smith group
Drug: Propofol — Manual control group: Propofol administration adjusted manually.
  Arms: 1: Manual control group

SUMMARY:
The action of anesthetics such as propofol is not immediate after intravenous administration. Delay in pharmacodynamic effect of intravenous drugs is a commonly observed phenomenon in total intravenous anesthesia (TIVA). On the other hand, the measure of the clinical effect of propofol by EEG processed monitors like the bispectral index (BIS) also requires some processing time for the analysis of the recorded signal. Thus, the resulting BIS value provided by the monitor is affected by a delay. When a BIS based controller is used, the propofol infusion rates are defined using information of the BIS signal available. The delay in the BIS signal is an important issue as it can affect the performance of the controller. There are scarce contributions to address the delay in automatic administration of anesthesia.

Our proposal to deal with the dead time in the control action of the hypnotic component of anesthesia is a proportional-integral (PI) algorithm with a Smith predictor. The aim of this study is to evaluate and compare the feasibility and effectiveness of a closed-loop control using the Smith predictor versus manual control for propofol administration guided by the bispectral index (BIS) in adults patients. The objective is to show that a closed loop control can be a useful tool to provide safe and effective intravenous anesthesia and that the use of specific controller for delay rejection is a reliable strategy.

DETAILED DESCRIPTION:
Modern medicine is focused on individualized treatment, including a personalized anesthesia administration. This implies to maintain the patient hypnotic state as closer as possible to a set target. TIVA with propofol and remifentanil has increased in popularity in recent years. Automatic systems can free the anesthesiologist of repetitive tasks. So, closed loop administration has been proposed to adjust propofol infusion rate without anesthesiologist intervention apart from supervising the procedure. A desired target of BIS is chosen by the clinician and feedback from the BIS monitor is used to adjust the rate of drug delivery continuously.

Closed loop control offers the opportunity of adjust the administration of anesthetics in an individualized way. It is also expected to overcome the individual pharmacokinetic and pharmacodynamic variability and to show a better adaptation to different levels of surgical stimulation. Closed loop control of propofol administration provides a greater stability in the level of hypnosis with a lower total dose of drug administered. Therefore, the recovery after anesthesia can be shorter. This can promote a better quality anesthetic care.

Previous studies with a PI controller showed in some patients a tendency to oscillate around a target value. This can be originated by the delay present in the system. One of the most known strategies in engineering to face the delay in closed loop is the Smith predictor. The purpose of this study is to evaluate and compare the feasibility and efficacy of a closed-loop control with a PI plus a Smith predictor algorithm versus manual control for propofol administration guided by the bispectral index (BIS) in adults patients.

Two groups of 25 adult patients scheduled for gynecological, urologic or abdominal surgery with an estimated duration > 30 minutes will be enrolled and randomized to one of the 2 groups. In the Manual control group (MC), the propofol infusion rate will be adjusted at the discretion of the anesthesiologist. In the PI+Smith group, propofol will be administered automatically by the closed-loop anesthesia system. The controller calculated automatically the error (target BIS - actual BIS) every 5 s and governed the infusion pump adapting the rate of propofol. The goal in both groups is to maintain BIS between 40 and 60 during maintenance phase of anesthesia. This is the recommended range of BIS for an adequate level of hypnosis during general anesthesia. Remifentanil will be infused for analgesia with the objective of to avoid an inadequate level of analgesia that could affect the stability of BIS signal.

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide informed consent
* 18 years of age or older
* Classification of the American Society of Anesthesiologists (ASA) as I or II
* Elective surgical procedures requiring general anesthesia with an estimated duration > 30 minutes

Exclusion Criteria:

* Pregnant women,
* Patients with neurological or psychiatric disorders
* Patients taking any medication known to influence the EEG and subsequently the BIS

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2017-03-06 (Estimated); Primary Completion 2017-09-15 (Estimated); Study Completion 2017-09-15 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the performance of the 2 groups with the global score (GS). | During anesthesia maintenance, approximately 9 hours
  Global score is a calculated parameter which gives an idea of the overall performance of a closed-loop system. It is calculated as the sum of MDAPE and wobble divided by the fraction of time BIS was within ±10 of the target. The target BIS chosen will be 50. The GS is calculated according the formula:
  GS = (MDAPE + wobble)/ % of time with BIS between 40 and 60

SECONDARY OUTCOMES:
The percentage of time with BIS values within +/10 % of target BIS. | During anesthesia maintenance, approximately 9 hours
  Adequate depth of anaesthesia during surgical interventions
MDPE (median performance error) | During anesthesia maintenance, approximately 9 hours
  The difference between the observed and target value of BIS.
MDAPE (median absolute performance error): | During anesthesia maintenance, approximately 9 hours
  The median of the absolute values of performance errors.
Wobble | During anesthesia maintenance, approximately 9 hours
  The median of the difference between individual PE and the MDPE for each participant, it measures the intra-individual variability of PE.
Time to eyes opening | 30 minutes after the end of the anesthesia
  Time from discontinuation of the propofol and remifentanil infusions until the patient is able to open his eyes on command.
Time to tracheal extubation: | 30 minutes after the end of the anesthesia
  Time from discontinuation of propofol infusion until endotracheal tube removal.
Total consumption of propofol and remifentanil during anesthesia maintenance | During anesthesia maintenance, approximately 9 hours
  Propofol administered

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitario de Canarias, San Cristóbal de La Laguna, Santa Cruz de Tenerife, Spain

IPD SHARING:
Plan to Share IPD: No